CLINICAL TRIAL: NCT00005267
Title: Family Blood Pressure Program - HyperGEN
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1151; 5R01HL055673-15 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2012-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tissue suitable for DNA extraction

SUMMARY:
To map and identify the major genetic determinants of hypertension and to study possible interactions between genetic and non-genetic factors in defined populations. HyperGEN initially consisted of a nine grant network, which in turn is part of an NHLBI initiative, the Family Blood Pressure Program (FBPP) consisting of four networks.

DETAILED DESCRIPTION:
BACKGROUND:

Hypertension, a complex disease involving the interplay of genetic and environmental factors, affects an estimated 50 million Americans and is a major predisposing factor for myocardial infarction, vascular disease, stroke, and renal failure. It has been estimated from segregation analysis and twin studies that approximately 45 percent of the interindividual differences in blood pressure are accounted for by genetic differences. The identification of the genes whose variants contribute to high blood pressure will have far-reaching effects on our understanding of the pathophysiology of the circulation and may suggest new preventive measures and rational therapeutic approaches.

One of the principal advantages of the genetic approach is that it identifies primary molecular defects. As a result, it will be possible to stratify the general hypertensive population into subgroups based on genotype and intermediate phenotype and thereby evaluate preventive strategies and therapeutic approaches in more homogeneous groups. In addition, the identification of hypertensive genes also provides the basis for an understanding of the interactions between genes and environmental factors. It is very likely that particular environmental variables exert their effects only in the presence of certain genotypes.

Until recently, the techniques for dissecting the genetic determinants of high blood pressure were not available or were not developed to an extent that would make the Family Blood Pressure Program initiative feasible. However, several recent advances in technology and analytical methods, together with the rapid construction of genetic maps, have substantially improved the chances of detecting these genetic factors.

The concept for the Family Blood Pressure Program was conceived in the Report of the Expert Panel on Genetic Strategies for Heart, Lung, and Blood Diseases. The initiative was approved by the Arteriosclerosis, Hypertension, and Lipid Metabolism Advisory Committee (AHLMAC) in March, 1993. The genetic-epidemiological aspects were approved by the Clinical Applications and Prevention Advisory Committee (CAPAC) in February, 1993. The Request for Applications was released in March, 1994. Awards were made in September, 1995.

DESIGN NARRATIVE:

The network consists of five field centers, a central biochemistry laboratory, a molecular genetics laboratory, and a data coordinating center to study an equal sample of Black and non-Black families with two or more hypertensive siblings, untreated relatives, and controls for genetic association and sib-sib linkage studies. The studies, using samples from the Family Heart Study (FHS) and the Atherosclerosis Risk in Communities (ARIC) study, include determination and characterization of genes promoting hypertension and interaction with non-genetic factors.

Beginning in 1996, Donna Arnett, principal investigator of the University of Minnesota echocardiographic center under R01HL55673 , is performing a targeted echocardiographic exam on 3,100 HyperGEN participants in five field centers as part of the HyperGEN clinical examination. She is examining the genetics of left ventricular hypertrophy. Her study characterizes left ventricular structure and function, defines left ventricular structural phenotypes based on four geometric patterns (normal geometry, concentric remodeling, concentric left ventricular hypertrophy, and eccentric left ventricular hypertrophy). She examines a highly select group of candidate genes and their association with left ventricular mass and geometric pattern. Using quantitative trait loci analyses, she is testing for linkage of 240 anonymous, evenly spaced genetic markers with left ventricular mass and geometric patterns. She is also evaluating interactions between genes and potential risk factors for left ventricular hypertrophy, including insulin, glucose, blood pressure response to mental and physical stressors, dietary and urinary electrolytes, and obesity. The grant was not part of the original initiative. Approximately $2,093,000 support will be provided for this grant, broken down as follows: FY 1996 - $652,085; FY 1997 - $628,979; FY 1998 - $433,000; FY 1999 - $379,000.

The Family Blood Pressure Program, including HyperGEN, was renewed in FY 2000. The Family Blood Pressure Program as a whole carried out five specific aims in the renewal period. These aims were grouped according to two complementary themes: First, the investigators created and analyzed a database of blood pressure-related phenotype and genotype data from all FBPP participants (Aim 1). Within linked regions, they identified allelic variation within positional candidate genes and evaluated the relationship of these polymorphisms with blood pressure levels and hypertension status (Aims 2 and 3). Second, they used quantitative measures of target organ damage to identify genes that influence susceptibility to develop hypertensive heart and kidney diseases (Aims 4 and 5). In addition to the Program specific aims, each network, including HyperGEN, carried out its own specific aims alone, based on unique aspects of their population and interests and expertise of the investigators.

The HyperGEN network has taken the lead in studying associated subphenotypes of hypertension and will study the following: measures of metabolic intermediates such as plasma insulin, glucose and lipid levels, and red cell sodium-lithium transport; co-morbidity with diseases of possible common etiology such as diabetes, obesity, and hypertension-associated kidney disease; degree of specific target organ damage; differential response to environmental input; and left ventricular hypertrophy and other phenotypes measured by echocardiography. Co-morbid conditions and measures of end-organ damage will be used as stratifying variables. Genes that influence variation in measures of metabolic intermediates, blood pressure response to stressors, and left ventricular hypertrophy will be studied in linkage and association studies. Environmental exposures (medication use, activity level, smoking) will be used as covariates. These measurements will allow for the identification of genes that influence variation in these subphenotypes, some of which may overlap with genes that influence blood pressure levels per se, and others which may be specific to the associated phenotype, nearly all of which have heritabilities equivalent to or greater than blood pressure by itself.

The HyperGen was extended through August, 2008 to make the Program a shared resource for hypertension researchers in the United States and throughout the world. In Aim 1, the investigators will build, maintain and update a publicly available knowledge-base to facilitate research by non-FBPP investigators on the genetics of hypertension, its risk factors and its complications. In Aim 2, they will use state-of-the-art genetic linkage analysis methods to identify additional linkage regions using subgroups of pedigrees and physiologically relevant combinations of phenotypes that will aid in localizing hypertension genes. In Aim 3, they will use a combination of bioinformatics, a dense array of SNPs, and state-of-the-art data analysis to follow-up regions of interest and identify the underlying hypertension genes. The regions to be followed-up include those identified during the current phase of the FBPP and Aim 2 of this renewal phase. In Aim 4, they will evaluate the hypertension genes identified in Aim 3 for their association with multiple measures reflecting the cardiovascular and renal complications of hypertension, including left ventricular mass and microalbuminuria. It is the long-term goal of the FBPP to have the hypertension genetics community develop a comprehensive picture of the genetic architecture of human hypertension, including its risk factors, complications, and response to treatment.

ELIGIBILITY:
Inclusion criteria for probands: Onset of hypertension by age 60 years and the presence of at least one additional hypertensive sibling who was willing to participate. Hypertension was defined according to systolic BP ≥140 or diastolic BP ≥90 in at least two different evaluations, or treatment for hypertension. Volunteers with type 1 diabetes or renal failure were excluded.

Inclusion criteria for subsequent recruits: Criteria as indicated in Study Population Description (i.e., criteria based on familial relationships, hypertension and antihypertensive medication status).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: (A) sample of hypertensive sibships with at least two members diagnosed with hypertension before the age of 60 (probands); (B) random sample of age-matched persons from the same base populations, from which normotensive controls could be drawn; (C) unmedicated, normotensive adult offspring of one of the hypertensive siblings.
Sampling Method: Non-Probability Sample
Enrollment: 3604 (Actual)
Dates: Start 1995-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Arnett, Principal Investigator — University of Alabama at Birmingham; John Eckfeldt, Principal Investigator — University of Minnesota; R.Curtis Ellison, Principal Investigator — Boston University; Steven Hunt, Principal Investigator — University of Utah; Jean-Marc Lalouel, Principal Investigator — University of Utah; Cora Lewis, Principal Investigator — University of Alabama at Birmingham; Kari North, Principal Investigator — University of North Carolina; James Pankow, Principal Investigator — University of Minnesota; Dabeeru Rao, Principal Investigator — Washington University School of Medicine

REFERENCES:
- [Background] Province MA, Boerwinkle E, Chakravarti A, Cooper R, Fornage M, Leppert M, Risch N, Ranade K. Lack of association of the angiotensinogen-6 polymorphism with blood pressure levels in the comprehensive NHLBI Family Blood Pressure Program. National Heart, Lung and Blood Institute. J Hypertens. 2000 Jul;18(7):867-76. doi: 10.1097/00004872-200018070-00008. PMID 10930184
- [Background] Williams RR, Rao DC, Ellison RC, Arnett DK, Heiss G, Oberman A, Eckfeldt JH, Leppert MF, Province MA, Mockrin SC, Hunt SC. NHLBI family blood pressure program: methodology and recruitment in the HyperGEN network. Hypertension genetic epidemiology network. Ann Epidemiol. 2000 Aug;10(6):389-400. doi: 10.1016/s1047-2797(00)00063-6. PMID 10964005
- [Background] Province MA, Arnett DK, Hunt SC, Leiendecker-Foster C, Eckfeldt JH, Oberman A, Ellison RC, Heiss G, Mockrin SC, Williams RR. Association between the alpha-adducin gene and hypertension in the HyperGEN Study. Am J Hypertens. 2000 Jun;13(6 Pt 1):710-8. doi: 10.1016/s0895-7061(99)00282-4. PMID 10912758
- [Background] Province MA. Sequential methods of analysis for genome scans. Adv Genet. 2001;42:499-514. doi: 10.1016/s0065-2660(01)42039-6. PMID 11037338
- [Background] Palmieri V, Bella JN, Arnett DK, Liu JE, Oberman A, Schuck MY, Kitzman DW, Hopkins PN, Morgan D, Rao DC, Devereux RB. Effect of type 2 diabetes mellitus on left ventricular geometry and systolic function in hypertensive subjects: Hypertension Genetic Epidemiology Network (HyperGEN) study. Circulation. 2001 Jan 2;103(1):102-7. doi: 10.1161/01.cir.103.1.102. PMID 11136693
- [Background] DeWan AT, Arnett DK, Atwood LD, Province MA, Lewis CE, Hunt SC, Eckfeldt J. A genome scan for renal function among hypertensives: the HyperGEN study. Am J Hum Genet. 2001 Jan;68(1):136-144. doi: 10.1086/316927. Epub 2000 Dec 12. PMID 11115379
- [Background] de Simone G, Palmieri V, Bella JN, Celentano A, Hong Y, Oberman A, Kitzman DW, Hopkins PN, Arnett DK, Devereux RB. Association of left ventricular hypertrophy with metabolic risk factors: the HyperGEN study. J Hypertens. 2002 Feb;20(2):323-31. doi: 10.1097/00004872-200202000-00024. PMID 11821719
- [Background] Arnett DK, Hong Y, Bella JN, Oberman A, Kitzman DW, Hopkins PN, Rao DC, Devereux RB. Sibling correlation of left ventricular mass and geometry in hypertensive African Americans and whites: the HyperGEN study. Hypertension Genetic Epidemiology Network. Am J Hypertens. 2001 Dec;14(12):1226-30. doi: 10.1016/s0895-7061(01)02200-2. PMID 11775131
- [Background] Arnett DK, Devereux RB, Kitzman D, Oberman A, Hopkins P, Atwood L, Dewan A, Rao DC; Hypertension Genetic Epidemiology Network Study Group. Linkage of left ventricular contractility to chromosome 11 in humans: The HyperGEN Study. Hypertension. 2001 Oct;38(4):767-72. doi: 10.1161/hy1001.092650. PMID 11641284
- [Background] Bella JN, Palmieri V, Liu JE, Kitzman DW, Oberman A, Hunt SC, Hopkins PN, Rao DC, Arnett DK, Devereux RB; Hypertension Genetic Epidemiology Network Study Group. Relationship between left ventricular diastolic relaxation and systolic function in hypertension: The Hypertension Genetic Epidemiology Network (HyperGEN) Study. Hypertension. 2001 Sep;38(3):424-8. doi: 10.1161/01.hyp.38.3.424. PMID 11566916
- [Background] Devereux RB, Bella JN, Palmieri V, Oberman A, Kitzman DW, Hopkins PN, Rao DC, Morgan D, Paranicas M, Fishman D, Arnett DK; Hypertension Genetic Epidemiology Network Study Group. Left ventricular systolic dysfunction in a biracial sample of hypertensive adults: The Hypertension Genetic Epidemiology Network (HyperGEN) Study. Hypertension. 2001 Sep;38(3):417-23. doi: 10.1161/01.hyp.38.3.417. PMID 11566915
- [Background] Palmieri V, Bella JN, Arnett DK, Roman MJ, Oberman A, Kitzman DW, Hopkins PN, Paranicas M, Rao DC, Devereux RB. Aortic root dilatation at sinuses of valsalva and aortic regurgitation in hypertensive and normotensive subjects: The Hypertension Genetic Epidemiology Network Study. Hypertension. 2001 May;37(5):1229-35. doi: 10.1161/01.hyp.37.5.1229. PMID 11358933
- [Background] Wu X, Cooper RS, Borecki I, Hanis C, Bray M, Lewis CE, Zhu X, Kan D, Luke A, Curb D. A combined analysis of genomewide linkage scans for body mass index from the National Heart, Lung, and Blood Institute Family Blood Pressure Program. Am J Hum Genet. 2002 May;70(5):1247-56. doi: 10.1086/340362. Epub 2002 Mar 28. PMID 11923912
- [Background] Coon H, Leppert MF, Eckfeldt JH, Oberman A, Myers RH, Peacock JM, Province MA, Hopkins PN, Heiss G. Genome-wide linkage analysis of lipids in the Hypertension Genetic Epidemiology Network (HyperGEN) Blood Pressure Study. Arterioscler Thromb Vasc Biol. 2001 Dec;21(12):1969-76. doi: 10.1161/hq1201.100228. PMID 11742872
- [Background] Palmieri V, de Simone G, Arnett DK, Bella JN, Kitzman DW, Oberman A, Hopkins PN, Province MA, Devereux RB. Relation of various degrees of body mass index in patients with systemic hypertension to left ventricular mass, cardiac output, and peripheral resistance (The Hypertension Genetic Epidemiology Network Study). Am J Cardiol. 2001 Nov 15;88(10):1163-8. doi: 10.1016/s0002-9149(01)02054-9. PMID 11703964
- [Background] Bella JN, Palmieri V, Kitzman DW, Liu JE, Oberman A, Hunt SC, Hopkins PN, Rao DC, Arnett DK, Devereux RB. Gender difference in diastolic function in hypertension (the HyperGEN study). Am J Cardiol. 2002 May 1;89(9):1052-6. doi: 10.1016/s0002-9149(02)02274-9. PMID 11988194
- [Background] Tang W, Devereux RB, Rao DC, Oberman A, Hopkins PN, Kitzman DW, Arnett DK. Associations between angiotensinogen gene variants and left ventricular mass and function in the HyperGEN study. Am Heart J. 2002 May;143(5):854-60. doi: 10.1067/mhj.2002.121926. PMID 12040348
- [Background] Palmieri V, Arnett DK, Roman MJ, Liu JE, Bella JN, Oberman A, Kitzman DW, Hopkins PN, Morgan D, de Simone G, Devereux RB. Appetite suppressants and valvular heart disease in a population-based sample: the HyperGEN study. Am J Med. 2002 Jun 15;112(9):710-5. doi: 10.1016/s0002-9343(02)01123-3. PMID 12079711
- [Background] Tang W, Arnett DK, Devereux RB, Atwood LD, Kitzman DW, Rao DC. Linkage of left ventricular early diastolic peak filling velocity to chromosome 5 in hypertensive African Americans: the HyperGEN echocardiography study. Am J Hypertens. 2002 Jul;15(7 Pt 1):621-7. doi: 10.1016/s0895-7061(02)02943-6. PMID 12118910
- [Background] Wilk JB, Myers RH, Zhang Y, Lewis CE, Atwood L, Hopkins PN, Ellison RC. Evidence for a gene influencing heart rate on chromosome 4 among hypertensives. Hum Genet. 2002 Aug;111(2):207-13. doi: 10.1007/s00439-002-0780-9. Epub 2002 Jul 16. PMID 12189495
- [Background] Devereux RB, de Simone G, Palmieri V, Oberman A, Hopkins P, Kitzman DW, Rao DC, Arnett DK. Relation of insulin to left ventricular geometry and function in African American and white hypertensive adults: the HyperGEN study. Am J Hypertens. 2002 Dec;15(12):1029-35. doi: 10.1016/s0895-7061(02)03080-7. PMID 12460697
- [Background] al'Absi M, Devereux RB, Lewis CE, Kitzman DW, Rao DC, Hopkins P, Markovitz J, Arnett DK. Blood pressure responses to acute stress and left ventricular mass (The Hypertension Genetic Epidemiology Network Study). Am J Cardiol. 2002 Mar 1;89(5):536-40. doi: 10.1016/s0002-9149(01)02305-0. PMID 11867037
- [Background] Tang W, Arnett DK, Devereux RB, Province MA, Atwood LD, Oberman A, Hopkins PN, Kitzman DW. Sibling resemblance for left ventricular structure, contractility, and diastolic filling. Hypertension. 2002 Sep;40(3):233-8. doi: 10.1161/01.hyp.0000028487.62501.12. PMID 12215459
- [Background] DeWan AT, Arnett DK, Miller MB, Peacock JM, Atwood LD, Province MA, Lewis CE, Hunt SC, Eckfeldt JH. Refined mapping of suggestive linkage to renal function in African Americans: the HyperGEN study. Am J Hum Genet. 2002 Jul;71(1):204-5. doi: 10.1086/340730. No abstract available. PMID 12068377
- [Background] Province MA, Kardia SL, Ranade K, Rao DC, Thiel BA, Cooper RS, Risch N, Turner ST, Cox DR, Hunt SC, Weder AB, Boerwinkle E; National Heart, Lung and Blood Institute Family Blood Pressure Program. A meta-analysis of genome-wide linkage scans for hypertension: the National Heart, Lung and Blood Institute Family Blood Pressure Program. Am J Hypertens. 2003 Feb;16(2):144-7. doi: 10.1016/s0895-7061(02)03248-x. PMID 12559682
- [Background] Rao DC, Province MA, Leppert MF, Oberman Al, Heiss G, Ellison RC, Arnett DK, Eckfeldt JH, Schwander K, Mockrin SC, Hunt SC; HyperGEN Network. A genome-wide affected sibpair linkage analysis of hypertension: the HyperGEN network. Am J Hypertens. 2003 Feb;16(2):148-50. doi: 10.1016/s0895-7061(02)03247-8. PMID 12559683
- [Background] Palmieri V, Bella JN, Arnett DK, Oberman A, Kitzman DW, Hopkins PN, Rao DC, Roman MJ, Devereux RB; Hypertension Genetic Epidemiology Network study. Associations of aortic and mitral regurgitation with body composition and myocardial energy expenditure in adults with hypertension: the Hypertension Genetic Epidemiology Network study. Am Heart J. 2003 Jun;145(6):1071-7. doi: 10.1016/S0002-8703(03)00099-1. PMID 12796765
- [Background] Freedman BI, Beck SR, Rich SS, Heiss G, Lewis CE, Turner S, Province MA, Schwander KL, Arnett DK, Mellen BG; HyperGEN Investigators. A genome-wide scan for urinary albumin excretion in hypertensive families. Hypertension. 2003 Sep;42(3):291-6. doi: 10.1161/01.HYP.0000087890.33245.41. Epub 2003 Aug 18. PMID 12925555
- [Background] de Simone G, Devereux RB, Palmieri V, Bella JN, Oberman A, Kitzman DW, Hopkins PN, Rao DC, Arnett DK; HyperGEN Study. Influence of fat-free mass on detection of appropriateness of left ventricular mass: the HyperGEN Study. J Hypertens. 2003 Sep;21(9):1747-52. doi: 10.1097/00004872-200309000-00025. PMID 12923408
- [Background] Kizer JR, Arnett DK, Bella JN, Paranicas M, Rao DC, Province MA, Oberman A, Kitzman DW, Hopkins PN, Liu JE, Devereux RB. Differences in left ventricular structure between black and white hypertensive adults: the Hypertension Genetic Epidemiology Network study. Hypertension. 2004 Jun;43(6):1182-8. doi: 10.1161/01.HYP.0000128738.94190.9f. Epub 2004 May 3. PMID 15123573
- [Background] Barkley RA, Chakravarti A, Cooper RS, Ellison RC, Hunt SC, Province MA, Turner ST, Weder AB, Boerwinkle E; Family Blood Pressure Program. Positional identification of hypertension susceptibility genes on chromosome 2. Hypertension. 2004 Feb;43(2):477-82. doi: 10.1161/01.HYP.0000111585.76299.f7. Epub 2004 Jan 19. PMID 14732741
- [Background] de Simone G, Kitzman DW, Palmieri V, Liu JE, Oberman A, Hopkins PN, Bella JN, Rao DC, Arnett DK, Devereux RB. Association of inappropriate left ventricular mass with systolic and diastolic dysfunction: the HyperGEN study. Am J Hypertens. 2004 Sep;17(9):828-33. doi: 10.1016/j.amjhyper.2004.04.008. PMID 15363827
- [Background] Wilk JB, Djousse L, Arnett DK, Hunt SC, Province MA, Heiss G, Myers RH. Genome-wide linkage analyses for age at diagnosis of hypertension and early-onset hypertension in the HyperGEN study. Am J Hypertens. 2004 Sep;17(9):839-44. doi: 10.1016/j.amjhyper.2004.06.003. PMID 15363829
- [Background] Morrison AC, Cooper R, Hunt S, Lewis CE, Luke A, Mosley TH, Boerwinkle E. Genome scan for hypertension in nonobese African Americans: the National Heart, Lung, and Blood Institute Family Blood Pressure Program. Am J Hypertens. 2004 Sep;17(9):834-8. doi: 10.1016/j.amjhyper.2004.04.009. PMID 15363828
- [Background] Kraja AT, Hunt SC, Pankow JS, Myers RH, Heiss G, Lewis CE, Rao D, Province MA. An evaluation of the metabolic syndrome in the HyperGEN study. Nutr Metab (Lond). 2005 Jan 18;2(1):2. doi: 10.1186/1743-7075-2-2. PMID 15656912
- [Background] de Simone G, Kitzman DW, Chinali M, Oberman A, Hopkins PN, Rao DC, Arnett DK, Devereux RB. Left ventricular concentric geometry is associated with impaired relaxation in hypertension: the HyperGEN study. Eur Heart J. 2005 May;26(10):1039-45. doi: 10.1093/eurheartj/ehi019. Epub 2004 Nov 30. PMID 15618056
- [Background] North KE, Rose KM, Borecki IB, Oberman A, Hunt SC, Miller MB, Blangero J, Almasy L, Pankow JS. Evidence for a gene on chromosome 13 influencing postural systolic blood pressure change and body mass index. Hypertension. 2004 Apr;43(4):780-4. doi: 10.1161/01.HYP.0000118921.66329.da. Epub 2004 Feb 16. PMID 14967843
- [Background] Tang H, Quertermous T, Rodriguez B, Kardia SL, Zhu X, Brown A, Pankow JS, Province MA, Hunt SC, Boerwinkle E, Schork NJ, Risch NJ. Genetic structure, self-identified race/ethnicity, and confounding in case-control association studies. Am J Hum Genet. 2005 Feb;76(2):268-75. doi: 10.1086/427888. Epub 2004 Dec 29. PMID 15625622
- [Background] Avery CL, Freedman BI, Heiss G, Kraja A, Rice T, Arnett D, Miller MB, Pankow JS, Lewis CE, Myers RH, Hunt SC, Almasy L, North KE; Hypertension Genetic Epidemiology Network. Linkage analysis of diabetes status among hypertensive families: the Hypertension Genetic Epidemiology Network study. Diabetes. 2004 Dec;53(12):3307-12. doi: 10.2337/diabetes.53.12.3307. PMID 15561964
- [Background] Freedman BI, Rich SS, Sale MM, Heiss G, Djousse L, Pankow JS, Province MA, Rao DC, Lewis CE, Chen YD, Beck SR; HyperGEN Investigators. Genome-wide scans for heritability of fasting serum insulin and glucose concentrations in hypertensive families. Diabetologia. 2005 Apr;48(4):661-8. doi: 10.1007/s00125-005-1679-5. Epub 2005 Mar 4. PMID 15747111
- [Background] An P, Freedman BI, Hanis CL, Chen YD, Weder AB, Schork NJ, Boerwinkle E, Province MA, Hsiung CA, Wu X, Quertermous T, Rao DC. Genome-wide linkage scans for fasting glucose, insulin, and insulin resistance in the National Heart, Lung, and Blood Institute Family Blood Pressure Program: evidence of linkages to chromosome 7q36 and 19q13 from meta-analysis. Diabetes. 2005 Mar;54(3):909-14. doi: 10.2337/diabetes.54.3.909. PMID 15734873
- [Background] Zhu X, Luke A, Cooper RS, Quertermous T, Hanis C, Mosley T, Gu CC, Tang H, Rao DC, Risch N, Weder A. Admixture mapping for hypertension loci with genome-scan markers. Nat Genet. 2005 Feb;37(2):177-81. doi: 10.1038/ng1510. Epub 2005 Jan 23. PMID 15665825
- [Background] Jorgenson E, Tang H, Gadde M, Province M, Leppert M, Kardia S, Schork N, Cooper R, Rao DC, Boerwinkle E, Risch N. Ethnicity and human genetic linkage maps. Am J Hum Genet. 2005 Feb;76(2):276-90. doi: 10.1086/427926. Epub 2004 Dec 30. PMID 15627237
- [Background] de Simone G, Devereux RB, Kizer JR, Chinali M, Bella JN, Oberman A, Kitzman DW, Hopkins PN, Rao DC, Arnett DK. Body composition and fat distribution influence systemic hemodynamics in the absence of obesity: the HyperGEN Study. Am J Clin Nutr. 2005 Apr;81(4):757-61. doi: 10.1093/ajcn/81.4.757. PMID 15817849
- [Background] Pankow JS, Dunn DM, Hunt SC, Leppert MF, Miller MB, Rao DC, Heiss G, Oberman A, Lalouel JM, Weiss RB. Further evidence of a quantitative trait locus on chromosome 18 influencing postural change in systolic blood pressure: the Hypertension Genetic Epidemiology Network (HyperGEN) Study. Am J Hypertens. 2005 May;18(5 Pt 1):672-8. doi: 10.1016/j.amjhyper.2004.12.004. PMID 15882550
- [Background] Lynch AI, Arnett DK, Atwood LD, Devereux RB, Kitzman DW, Hopkins PN, Oberman A, Rao DC. A genome scan for linkage with aortic root diameter in hypertensive African Americans and whites in the Hypertension Genetic Epidemiology Network (HyperGEN) study. Am J Hypertens. 2005 May;18(5 Pt 1):627-32. doi: 10.1016/j.amjhyper.2004.11.029. PMID 15882545
- [Background] Lewis CE, North KE, Arnett D, Borecki IB, Coon H, Ellison RC, Hunt SC, Oberman A, Rich SS, Province MA, Miller MB. Sex-specific findings from a genome-wide linkage analysis of human fatness in non-Hispanic whites and African Americans: the HyperGEN study. Int J Obes (Lond). 2005 Jun;29(6):639-49. doi: 10.1038/sj.ijo.0802916. PMID 15809668
- [Background] North KE, Miller MB, Coon H, Martin LJ, Peacock JM, Arnett D, Zhang B, Province M, Oberman A, Blangero J, Almasy L, Ellison RC, Heiss G. Evidence for a gene influencing fasting LDL cholesterol and triglyceride levels on chromosome 21q. Atherosclerosis. 2005 Mar;179(1):119-25. doi: 10.1016/j.atherosclerosis.2004.09.009. Epub 2004 Nov 14. PMID 15721017
- [Background] Agno FS, Chinali M, Bella JN, Liu JE, Arnett DK, Kitzman DW, Oberman A, Hopkins PN, Rao DC, Devereux RB. Aortic valve sclerosis is associated with preclinical cardiovascular disease in hypertensive adults: the Hypertension Genetic Epidemiology Network study. J Hypertens. 2005 Apr;23(4):867-73. doi: 10.1097/01.hjh.0000163157.14493.c7. PMID 15775793
- [Background] Arnett DK, Tang W, Province MA, Oberman A, Ellison RC, Morgan D, Eckfeldt JH, Hunt SC. Interarm differences in seated systolic and diastolic blood pressure: the Hypertension Genetic Epidemiology Network study. J Hypertens. 2005 Jun;23(6):1141-7. doi: 10.1097/01.hjh.0000170376.23461.f7. PMID 15894889
- [Background] Chinali M, de Simone G, Liu JE, Bella JN, Oberman A, Hopkins PN, Kitzman DW, Rao DC, Arnett DK, Devereux RB. Left atrial systolic force and cardiac markers of preclinical disease in hypertensive patients: the Hypertension Genetic Epidemiology Network (HyperGEN) Study. Am J Hypertens. 2005 Jul;18(7):899-905. doi: 10.1016/j.amjhyper.2005.01.005. PMID 16053984
- [Background] Kraja AT, Rao DC, Weder AB, Mosley TH, Turner ST, Hsiung CA, Quertermous T, Cooper R, Curb JD, Province MA. An evaluation of the metabolic syndrome in a large multi-ethnic study: the Family Blood Pressure Program. Nutr Metab (Lond). 2005 Aug 2;2:17. doi: 10.1186/1743-7075-2-17. PMID 16076393
- [Background] Kraja AT, Hunt SC, Pankow JS, Myers RH, Heiss G, Lewis CE, Rao DC, Province MA. Quantitative trait loci for metabolic syndrome in the Hypertension Genetic Epidemiology Network study. Obes Res. 2005 Nov;13(11):1885-90. doi: 10.1038/oby.2005.231. PMID 16339118
- [Background] Bielinski SJ, Lynch AI, Miller MB, Weder A, Cooper R, Oberman A, Chen YD, Turner ST, Fornage M, Province M, Arnett DK. Genome-wide linkage analysis for loci affecting pulse pressure: the Family Blood Pressure Program. Hypertension. 2005 Dec;46(6):1286-93. doi: 10.1161/01.HYP.0000191706.41980.29. Epub 2005 Nov 14. PMID 16286574
- [Derived] Li W, Turner A, Aggarwal P, Matter A, Storvick E, Arnett DK, Broeckel U. Comprehensive evaluation of AmpliSeq transcriptome, a novel targeted whole transcriptome RNA sequencing methodology for global gene expression analysis. BMC Genomics. 2015 Dec 16;16:1069. doi: 10.1186/s12864-015-2270-1. PMID 26673413
- [Derived] Scantlebury DC, Kane GC, Wiste HJ, Bailey KR, Turner ST, Arnett DK, Devereux RB, Mosley TH Jr, Hunt SC, Weder AB, Rodriguez B, Boerwinkle E, Weissgerber TL, Garovic VD. Left ventricular hypertrophy after hypertensive pregnancy disorders. Heart. 2015 Oct;101(19):1584-90. doi: 10.1136/heartjnl-2015-308098. Epub 2015 Aug 4. PMID 26243788
- [Derived] Glasser SP, Lynch AI, Devereux RB, Hopkins P, Arnett DK. Hemodynamic and echocardiographic profiles in African American compared with White offspring of hypertensive parents: the HyperGEN study. Am J Hypertens. 2014 Jan;27(1):21-6. doi: 10.1093/ajh/hpt178. Epub 2013 Nov 16. PMID 24242823
- [Derived] Liu CT, Monda KL, Taylor KC, Lange L, Demerath EW, Palmas W, Wojczynski MK, Ellis JC, Vitolins MZ, Liu S, Papanicolaou GJ, Irvin MR, Xue L, Griffin PJ, Nalls MA, Adeyemo A, Liu J, Li G, Ruiz-Narvaez EA, Chen WM, Chen F, Henderson BE, Millikan RC, Ambrosone CB, Strom SS, Guo X, Andrews JS, Sun YV, Mosley TH, Yanek LR, Shriner D, Haritunians T, Rotter JI, Speliotes EK, Smith M, Rosenberg L, Mychaleckyj J, Nayak U, Spruill I, Garvey WT, Pettaway C, Nyante S, Bandera EV, Britton AF, Zonderman AB, Rasmussen-Torvik LJ, Chen YD, Ding J, Lohman K, Kritchevsky SB, Zhao W, Peyser PA, Kardia SL, Kabagambe E, Broeckel U, Chen G, Zhou J, Wassertheil-Smoller S, Neuhouser ML, Rampersaud E, Psaty B, Kooperberg C, Manson JE, Kuller LH, Ochs-Balcom HM, Johnson KC, Sucheston L, Ordovas JM, Palmer JR, Haiman CA, McKnight B, Howard BV, Becker DM, Bielak LF, Liu Y, Allison MA, Grant SF, Burke GL, Patel SR, Schreiner PJ, Borecki IB, Evans MK, Taylor H, Sale MM, Howard V, Carlson CS, Rotimi CN, Cushman M, Harris TB, Reiner AP, Cupples LA, North KE, Fox CS. Genome-wide association of body fat distribution in African ancestry populations suggests new loci. PLoS Genet. 2013;9(8):e1003681. doi: 10.1371/journal.pgen.1003681. Epub 2013 Aug 15. PMID 23966867
- [Derived] Arnett DK, Meyers KJ, Devereux RB, Tiwari HK, Gu CC, Vaughan LK, Perry RT, Patki A, Claas SA, Sun YV, Broeckel U, Kardia SL. Genetic variation in NCAM1 contributes to left ventricular wall thickness in hypertensive families. Circ Res. 2011 Feb 4;108(3):279-83. doi: 10.1161/CIRCRESAHA.110.239210. Epub 2011 Jan 6. PMID 21212386
- [Derived] Arnett DK, Devereux RB, Rao DC, Li N, Tang W, Kraemer R, Claas SA, Leon JM, Broeckel U. Novel genetic variants contributing to left ventricular hypertrophy: the HyperGEN study. J Hypertens. 2009 Aug;27(8):1585-93. doi: 10.1097/HJH.0b013e32832be612. PMID 19593212